CLINICAL TRIAL: NCT05671835
Title: REVERT-IPF: A Phase 2 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of TTI-101 in Participants With Idiopathic Pulmonary Fibrosis
Brief Title: Study of TTI-101 in Participants With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tvardi Therapeutics, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVD-101-003P
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; IPF; TTI-101
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — C188-9 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TTI-101 400 mg/day (Experimental): Participants will receive 400 mg/day of TTI-101 twice daily (BID) for 12 weeks.
  Interventions: Drug: TTI-101
- TTI-101 800 mg/day (Experimental): Participants will receive 800 mg/day of TTI-101 BID for 12 weeks.
  Interventions: Drug: TTI-101
- Placebo (Placebo Comparator): Participants will receive a matching placebo BID for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTI-101 — Orally via a tablet.
  Arms: TTI-101 400 mg/day; TTI-101 800 mg/day
Drug: Placebo — Orally via a tablet.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of oral daily administration of TTI-101 over a 12-week treatment duration in participants with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with IPF based on either the 2018 American Thoracic Society (ATS)/ European Respiratory Society (ERS)/ Japanese Respiratory Society (JRS)/ Latin American Thoracic Association (ALAT) International Diagnostic Guidelines or on the 2022 updated guidelines within 7 years prior to the date of informed consent.
2. Chest high-resolution computed tomography scan (HRCT) performed within 12 months prior to providing informed consent meeting requirements for IPF diagnosis based on 2018 or 2022 ATS/ERS/JRS/ALAT guidelines and confirmed by central review.
3. Greater than 40% of predicted forced vital capacity (FVC) and a ratio of forced expiratory volume in 1 second (FEV1)/FVC ≥0.7 measured pre-bronchodilator during screening confirmed by central review.
4. A predicted diffusing capacity of the lungs for carbon monoxide (DLCO) (hemoglobin [Hb] corrected) ≥25% during screening confirmed by central review.
5. Oxygen saturation (SpO2) ≥88% with up to 4L O2/min by pulse oximetry at rest.
6. If currently receiving nintedanib, dose must have been stable for ≥3 months prior to randomization. If participant has previously discontinued nintedanib, there is a 6-week washout period required before screening can begin.
7. Has a life expectancy of at least 12 months.

Exclusion Criteria:

1. Unresolved respiratory tract infection within 4 weeks (including coronavirus disease 2019 [COVID-19] infections) or an acute exacerbation of IPF within 3 months prior to screening.
2. Planned surgery during the study.
3. The investigator judges that there has been sustained improvement in the severity of IPF during the 12 months prior to screening, based on changes in FVC, DLCO, and/or HRCT scans of the chest.
4. History of other types of respiratory diseases including diseases or disorders of the airways, lung parenchyma, pleural space, mediastinum, diaphragm, or chest wall that, in the opinion of the investigator, would impact the primary protocol endpoint or ability to do pulmonary function tests (PFTs), or otherwise preclude participation in the study.
5. Likely to have lung transplantation during the study. Note: Participant may be on a lung transplant list if the investigator anticipates the participant will be able to complete the study prior to transplant.
6. Clinically relevant and uncontrolled cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorders that may interfere with the participant's ability to complete this study according to the investigator's judgment, or logistical challenges that, in the opinion of the investigator, preclude adequate participation in the study.
7. History or difficulty of swallowing, malabsorption, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the study drug.
8. Receiving steroids (excluding topical steroids) in excess of a mean of 10 mg/day of prednisolone or its equivalent within 2 weeks prior to randomization.
9. Received pirfenidone within 3 months prior to randomization.
10. Smoking or vaping of any kind within 3 months of screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with an Adverse Event (AE) | 16 weeks
  Incidence of AEs, including serious AEs assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) V.5.0. Clinically significant changes between baseline and postbaseline laboratory assessments, electrocardiograms, vital signs, and physical examinations will be recorded as AEs.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of TTI-101 | Day 1 to Week 12
Time of Maximum Observed Plasma Concentration (tmax) of TTI-101 | Day 1 to Week 12
Area Under the Plasma Concentration-time Curve Over a Dosing Interval (AUC[0-τ]) of TTI-101 | Day 1 to Week 12
Trough Plasma Concentration (Cτ) of TTI-101 | Day 1 to Week 12

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - The Kirklin Clinic of University of Alabama Birmingham Hospital, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - University of California Irvine (UCI) Health, Orange, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Saint Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - UHealth - University of Miami Health Systems, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tulane University School of Medicine, New Orleans, Louisiana
  - The Lung Research Center, Chesterfield, Missouri
  - New York University Langone Pulmonary and Critical Care Associates, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Pulmonix, Greensboro, North Carolina
  - Salem Chest Specialists, Winston-Salem, North Carolina
  - Saint Luke's University Hospital - Bethlehem, Bethlehem, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Baylor Scott & White Center for Advanced Heart & Lung Disease, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston (UT Health), Houston, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No